CLINICAL TRIAL: NCT06328231
Title: The Effect of Simple Swallowing Rehabilitation Training for Elderly Community Dwellers: A Preliminary Study
Brief Title: The Impact of Swallowing Intervention for Elderly Community Dwellers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Community elderly dysphagia
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic simple swallowing training (Experimental): The elderly individuals will be arranged to undergo a continuous three-week (21 days) duration of systematic simple swallowing training, with weekends off and training conducted only on weekdays, two sessions per day, each lasting 15 minutes. Each training session will be conducted approximately one hour prior to meals. Apart from this,we require participants to only engage in daily activities and avoid strenuous and dangerous behaviors
  Interventions: Behavioral: Systematic simple swallowing training
- Blank Group (No Intervention): This group received no intervention but were requested to do mild physical activities by themselves

INTERVENTIONS:
Behavioral: Systematic simple swallowing training — Systematic simple swallowing training includes the following:
  Warm-up: including joint activities, chest expansion exercise, etc., totally 5 minutes.
  Cognitive swallowing training: play video of food programs for five minutes. Lip training: Bounce the upper and lower lips to make a "bo" sound. 30-60 seconds.
  Tongue training: Do the upper, lower, left, and right four-directional movements of the tongue muscle. 30-60 seconds.
  Mandibular training: slowly open r mouth to the maximum, then slowly close it. 30-60 seconds.
  Soft palate training: Make the sounds of g, k, and h for 1-2 minutes. Cheek puffing training: Close lips tightly and puff cheeks. 30-60 seconds. Swallowing training: We require the elderly to swallow small amounts of water intermittently and forcefully for 2-5 times.
  Completing the above content in succession is called a round, and each training session includes 2-3 rounds. 2 sessions a day. Five days a week.
  Arms: Systematic simple swallowing training

SUMMARY:
The goal of this clinical trial is to explore the impact of systematic simple swallowing training on swallowing function and quality of life in community-dwelling elderly individuals (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of dysphagia among community-dwelling elderly individuals, and 2) the effects of systematic simple swallowing training on swallowing function and quality of life in community-dwelling elderly individuals with swallowing disorders. All participants are divided into 2 groups. The intervention group is required to undergo a continuous three-week (21 days) systematic simple swallowing training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 15-20 minutes each.

DETAILED DESCRIPTION:
The investigators have designed a simple and user-friendly swallowing rehabilitation training method called "systematic simple swallowing training" based on commonly used swallowing training techniques in the department of rehabilitation medicine and the prevalent pathological causes of swallowing disorders in the elderly. It has shown promising preliminary efficacy. The goal of this clinical trial is to explore the impact of systematic simple swallowing training on swallowing function and quality of life in community-dwelling elderly individuals (≥60 year old) with swallowing disorders. It primarily aims to address two key aspects: 1) the prevalence of dysphagia among community-dwelling elderly individuals, and 2) the effects of systematic simple swallowing training on swallowing function and quality of life in community-dwelling elderly individuals with swallowing disorders. All participants are divided into 2 groups. The intervention group is required to undergo a continuous three-week (21 days) systematic simple swallowing training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 15-20 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old.
* No hospitalization within the past six months.
* With clear consciousness and able to cooperate with questionnaires and training.
* The elderly people who voluntarily participate and agree to adhere until the end of the study.
* early dysphagia.

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Physical disability.
* Difficulty in mobility.
* Simultaneously receiving other therapies that might influence this study.
* Individuals with a gastrostomy.
* Abnormalities of the oral, pharyngeal, or esophageal structures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Gugging Swallowing Screen | day 1 and day 21
  The Gugging Swallowing Screen is used to assess dysphagia. The Screen consists of 10 items covering various aspects of swallowing, including oral and pharyngeal muscle function, oral sensation, tongue coordination, and more. The total scores range from 1 to 20, with lower scores indicating more severe dysphagia.

SECONDARY OUTCOMES:
Time consumed in eating | day 1 and day 21
  We require participants to eat a lunch according to their daily intake and habits, and count the time consumed
Swallowing-Related Quality of Life Questionnaire | day 1 and day 21
  The Swallowing-Related Quality of Life Questionnaire (SWAL-QOL) is a validated tool used to assess the impact of swallowing difficulties on quality of life. It is a 44-item questionnaire designed to measure the physical, emotional, and social domains of swallowing-related quality of life.The higher final scores indicate the better life quality. The total score will be converted into a standard percentage
Eating Assessment Tool-10 | day 1 and day 21
  Subjective perception of swallowing function was assessed using the Eating Assessment Tool-10 (EAT-10). The EAT-10 comprises 10 questions that assess various aspects of swallowing function. Each question is scored on a scale from 0 to 4, indicating the severity of swallowing difficulty, with 0 for no difficulty and 4 for severe difficulty. Participants could rate it based on the subjective perception. The total score on the EAT-10 ranges from 0 to 40, with higher scores indicating more severe swallowing disorders.
Maximum tongue pressure | day 1 and day 21
  Tongue pressure instruments were used for maximum tongue pressure. The device measured the maximum pressure between the subject's tongue and the palate.
Bite force | day 1 and day 21
  Bite force testers were used for bite force. All subjects were instructed to try their best to bite it with centric dental occlusion
Masticatory ability | day 1 and day 21
  participants were required to chew 2g of gummy jelly relaxedly for twenty seconds. Then, 10 mL of water was used for gargling. The chewing materials were discharged to a filtering net. The glucose amount that passed the net was recorded with a glucose sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Principal Investigator — Site Coordinator of United Medical Group
Locations (1):
- Railway Commu., Zhenzhou, China

IPD SHARING:
Plan to Share IPD: No